CLINICAL TRIAL: NCT02401204
Title: Bacterial Transmission Surveillance in Neonatal Intensive Care Unit: Transmission Dynamics and Drug Resistance Patterns
Brief Title: Bacterial Transmission Dynamics Study
Acronym: BTS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Queen Sirikit National Institute of Child Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: MODEL1402
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Bacterial Transmission Surveillance; Neonatal Intensive Care Unit; Drug Resistance
Keywords: Bacterial transmission; Surveillance; Neonatal; Drug Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool Tracheal suction swab Rectal swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neonates admitted to QSNICH NICU: All neonates admitted to the QSNICH NICU over a period of one year from March 2015 to March 2016 meeting the inclusion and exclusion criteria will be enrolled in the study. Readmitted neonates will be eligible to be enrolled again into the study.
  Interventions: Other: Longitudinal surveillance study

INTERVENTIONS:
Other: Longitudinal surveillance study — Regular specimens will be routinely collected as standard of practice.
  A rectal swab and stool specimen will be collected twice a week since first admission on NICU until discharge from NICU.
  If participant is intubated/ventilated, a throat swab will be collected.

SUMMARY:
Infections with multiply antibiotic-resistant bacteria represent a major cause of preventable morbidity and mortality amongst hospitalized neonates worldwide. In Southeast Asia, where antibiotic-resistance is a major problem, Gram-negative bacteria account for the majority of such infections. The most common pathogens are Acinetobacter spp., Pseudomonas aeruginosa, Enterobacter spp., Escherichia coli and Klebsiella pneumonia. The great majority of infections with these pathogens represent asymptomatic carriage, though in the absence of routine screening for asymptomatic carriage reliable estimates of the prevalence, rates of transmission between patients, and rates of importation from the community are lacking. Moreover, current understanding of the degree and manner in which different antibiotics act to select for such resistant organisms is rudimentary.

DETAILED DESCRIPTION:
Objectives: To quantify the prevalence of drug-resistant Gram-negative pathogens on admission to a neonatal intensive care unit and during subsequent days of hospital stay. To quantify rates of patient-to-patient transmission for key organisms, to characterize how patient antibiotic use impacts on the ward-level dynamics of such organisms.

Methods: All infants admitted to the unit over a period of one year for whom the parent/guardian gives informed consent will be included. In addition to routine demographic and clinical data for included patients, full patient-level data on antibiotic use within the ward will also be recorded. Carriage of resistant Gram-negative organisms will be determined though rectal swabs, tracheal aspirates (for ventilated patients) and stool samples taken on admission and at twice weekly intervals. Antibiotic-resistant Gram-negative bacteria will be cultured and their resistant patterns determined. Selected environmental surfaces will also be sampled to detect contamination with such organisms. For the most important organisms (Acinetobacter spp. and Klebsiella spp.) whole genome sequencing will be used in conjunction with Bayesian data augmentation techniques to determine transmission pathways and the impact of antibiotic use on the transmission and persistence of such organisms within the hospital ward.

ELIGIBILITY:
Inclusion Criteria:

* All neonates admitted to QSNICH NICU
* Parent/legal guardian gives written informed consent

Exclusion Criteria:

• There are no exclusion criteria for this study

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates up to one month old
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Number of neonates who acquired infection from each expected pathogens during admission in NICU unit. | During admission in NICU unit

CONTACTS AND LOCATIONS:
Overall Officials: Ben Cooper, Dr., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Queen Sirikit National Institute of Child Health, Ratchathewi, Bangkok, Thailand